CLINICAL TRIAL: NCT06664970
Title: Prospective, Multicenter Study on the Treatment of Myelodysplastic Neoplasms (MDS)/Myeloproliferative Neoplasms (MPN) Overlap Syndrome With Azacitidine or Ruxolitinib Combined With Selinexor
Brief Title: A Multicenter Study on the Treatment of MDS/MPN Overlap Syndrome With AZA or Rux Combined With Selinexor
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, PekingUMCH, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K6812
Record Dates: First submitted 2024-10-09; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: MDS
MeSH Terms: interventions — Azacitidine; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Azacitidine or Ruxolitinib combined with Selinexor (Experimental): Azacitidine or Ruxolitinib combined with Selinexor
  Interventions: Drug: Azacitidine or Ruxolitinib combined with Selinexor

INTERVENTIONS:
Drug: Azacitidine or Ruxolitinib combined with Selinexor — 1. The initial dose of Selinexor combined with Azacitidine for the treatment of MDS patients is 40mg QW, adjusted according to blood tests, with the highest dose ≤ 60mg QW.
     Azacitidine: The initial dose is 75 mg/m ², administered subcutaneously or intravenously, with a cycle of 1-7 days and 28 days until ineffective or intolerant.
  2. Selinexor combined with Ruxolitinib for the treatment of patients with MPN symptoms: Selinexor dose: 40mg QW; Adjust according to the blood count, with a maximum dose of ≤ 60mg QW.
  Initial dose of Ruxolitinib: platelet count>100 × 109/L before enrollment, initial dose is 15 mg BID; Platelets range from 50-100 × 109/L, with an initial dose of 10 mg BID. Until ineffective or intolerant.

SUMMARY:
This study is a prospective, multicenter, open label cohort study involving MDS/MPN patients. The enrolled patients have symptoms that require treatment, which are classified according to their clinical conditions as follows: those with MDS as the main manifestation are treated with Azacitidine combined with Selinexor; For those with MPN as the main manifestation, treatment with Selinexor combined with Ruxolitinib is used.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria of MDS/MPN (WHO 2022 edition)
2. Age ≥ 18 years old;
3. There are indications that require treatment, such as symptomatic anemia, decreased blood cells, splenomegaly, and constitutional symptoms;
4. ECOG score 0-2;
5. No stem cell transplantation plan within 6 months;
6. Liver function: Within 21 days before the start of treatment, total bilirubin<2 times the upper limit of normal (ULN), alanine aminotransferase (ALT)<2.5 times ULN;
7. Renal function: Within 21 days before the start of treatment, creatinine clearance rate ≥ 30 mL/min, calculated using Cockcroft and Gault formulas;
8. Patients receiving erythropoietin therapy or rituximab must be at a stable dosage and have stable transfusion therapy or hemoglobin levels within 8 weeks prior to entering the study.
9. Female patients with fertility must agree to the use of dual contraception methods and have a negative serum pregnancy test during screening. Male patients who have sexual intercourse with women with fertility must use effective barrier contraception methods.
10. Those who meet the requirements of the ethics committee and sign the informed consent form; Willing and able to comply with clinical visit and research related procedures.

Exclusion Criteria:

1. Those who have undergone major surgery within 4 weeks before the start of treatment,
2. those with severe liver and kidney dysfunction;
3. Patients who have undergone splenectomy in the past;
4. Patients with unstable cardiovascular function: symptomatic cardiac ischemia, uncontrolled significant conduction abnormalities, congestive heart failure (CHF) with NYHA functional class ≥ 3 or myocardial infarction within 6 months, unstable angina, unstable arrhythmia;
5. Uncontrolled active infections require systemic use of antibiotics, antiviral drugs, or antifungal drugs within one week prior to the first administration; Allow the use of prophylactic antibiotics.
6. Known active hepatitis A, B, or C infection; Or known to be positive for HCV RNA or HBsAg (HBV surface antigen); Known HIV seropositivity;
7. Patients with obvious gastrointestinal lesions or obstruction, or uncontrolled vomiting or diarrhea.
8. At baseline, peripheral neuropathy was ≥ grade 2 (within 21 days before the first day of the first cycle).
9. History of epileptic seizures, movement disorders, or cerebrovascular accidents (within 1 year before the first day of the first cycle)
10. Evidence of AML (≥ 20% of primitive cells in bone marrow or peripheral blood) according to WHO definition
11. Patients with other active malignant tumors
12. Pregnant and lactating women;
13. Fertility capable women or men who are unwilling to take effective contraceptive measures before the first dose/treatment, during the study period, and for at least 6 months after the last dose;
14. Patients without autonomous behavioral ability, such as psychiatric patients; Other situations deemed unsuitable for inclusion by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-11-06 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR at 6 months of treatment | 6 months
  ORR at 6 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Bing Han, Beijing, China

IPD SHARING:
Plan to Share IPD: No